CLINICAL TRIAL: NCT00176111
Title: Effects of Local Anesthetic or Saline Solution on Peripheral Nerve Stimulation - a Randomised, Double-Blind, Multicenter Study About the Stimulability of Anesthetized Nerves
Brief Title: Effects of Local Anesthetic or Saline Solution on Peripheral Nerve Stimulation - a Randomised Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Rechbergklinik Bretten (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: nervstim001
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-17 (Estimated); Status verified 2004-01

CONDITIONS: Percutaneous Electric Nerve Stimulation
Keywords: peripheral nerve stimulation; saline; local anesthestics; regional anesthestia; nerve damage

INTERVENTIONS:
Procedure: peripheral nerve stimulation (procedure)

SUMMARY:
In this study we want to examine the effect of a small amount of local anesthetic or saline solution on nerve conduction using a peripheral nerve stimulator.

DETAILED DESCRIPTION:
Using electrical nerve stimulation in performing peripheral nerve helps to control the needle position in relation to the nerve and therefore may increase the likelihood of a successful nerve block. Defining the minimal stimulating current accepted also may help to avoid direct contact between nerve and needle or accidental endoneural injection and subsequent nerve lesion.

In recent years there have been many reports where several nerves, parts thereof or plexuses have been anesthetised using a multiple injection approach. That is, nerves in close proximity of each other have been subsequently blocked after using a nerve stimulator to locate them.

It is not clear though, whether a nerve may already be partially anesthetised in this situation and whether that would impair the correct use of a peripheral nerve stimulator.

The aim of this study is to examine the excitability of a peripheral nerve after injecting a small amount of local anesthetic agent or saline solution into the proximity of the nerve.

ELIGIBILITY:
Inclusion Criteria:

ASA 1-2

Exclusion Criteria:

peripheral neuropathy, ASA >2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Kaiser, MD, Study Chair — Rechbergklinik Bretten
Locations (1):
- Rechbergklinik, Bretten, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Neuburger M, Gultlinger O, Ass B, Buttner J, Kaiser H. [Influence of blockades with local anesthetics on the stimulation ability of a nerve by peripheral nerve stimulation. Results of a randomized study]. Anaesthesist. 2005 Jun;54(6):575-7. doi: 10.1007/s00101-005-0824-3. German. PMID 15739091